CLINICAL TRIAL: NCT04091919
Title: Assessment of Left and Right Ventricular Strain and Strain Rate Before and After Percutaneous Closure of Atrial Septal Defects in Adults and Adolescents
Brief Title: Assessment of LV/RV S and SR Before and After Percutaneous Closure of ASDs
Status: Completed | Type: Observational
Sponsor: Ayman khairy Mohamed (Other)
Responsible Party: Sponsor-Investigator, Ayman khairy Mohamed, Clinical Professor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: LV/RV S and SR with ASD device
Record Dates: First submitted 2019-09-11; First posted 2019-09-17 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Atrial Septal Defect, Secundum Type
Keywords: Left and right ventricular global longitudinal strain; ASD device closure
MeSH Terms: conditions — Atrial Septal Defect, Secundum Type | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- ASD group: Isolated ostium Secundum ASD patients who are involving in this study have been already selected for intervention before the starting time of the study. The ASD patients who will be scheduled for transcatheter closure have either haemodynamically significant shunt fraction (Qp/Qs > 1.5) or echocardiographic signs of right heart dilation or RV volume overload and pulmonary hypertension related symptoms. 2-D TTE derived Tissue Doppler and Strain Imaging will be done for all patients at baseline, 24 hours and 1-3 month post-procedure. Correlation between the device size and echocardiographic variables will be performed. Comparison between the results of the 2D-TTE derived Strain Imaging procedures will be done between baseline data and those obtained one day after the procedure and at one month follow up.
  Interventions: Diagnostic Test: 2D- Transthoracic Echocardiography (TTE)
- Controlled group: Age matched controlled subjects without ASD
  Interventions: Diagnostic Test: 2D- Transthoracic Echocardiography (TTE)

INTERVENTIONS:
Diagnostic Test: 2D- Transthoracic Echocardiography (TTE) — 2D- Transthoracic Echocardiography (TTE) derived Tissue Doppler and Strain imaging

SUMMARY:
The effect of Atrial Septal Defect (ASD) closure by using larger devices on the improvement in biventricular function remains an area of active research. Therefore, the aim of the current study is to assess the degree of improvement in biventricular dimensions and function by using 2-Dimensional echocardiography derived Strain and Strain Rate and Tissue Doppler. Moreover, to identify the relationship between the left and right ventricular systolic and diastolic function and device size.

DETAILED DESCRIPTION:
In most echocardiographic studies, left ventricle (LV) systolic function was normal in the patients with ASD and only a few cases had a reduced LV ejection fraction with severe right ventricle (RV) volume overload. The device closure of ASD increases immediately the blood flow to the left ventricle and may unmask subtle abnormalities in systolic and diastolic function. Currently, clinical research in cardiac mechanics is moving from short- and long-axis LV and RV function and ejection fraction to two and three- dimensional (2D, 3D) ventricular deformation studies (Strain and Strain Rate quantiﬁcation). These methods are independent of ventricular geometry and allow quantiﬁcation of myocardial motion and deformation in different directions (longitudinal, radial, and circumferential), while conventional methods mainly rely on the assessment of radial function. Strain imaging has also been used to demonstrate that patients who underwent device closure of an ASD had better LV and RV longitudinal deformation than patients who underwent surgical closure of an ASD. However, the effect of device size on the LV systolic and diastolic function is still under investigations. For all these reasons the researchers intend to measure RV and LV haemodynamic changes by 2-D Transthoracic Echocardiography (TTE) derived Tissue Doppler and Strain quantification in ASD before and after transcatheter closure with special emphasis on the assessment of the relationship between device size and biventricular systolic and LV diastolic function.

ELIGIBILITY:
Inclusion Criteria:

* All ASD patients who have been already selected and suitable for intervention before the starting time of the study. The criteria for ASD intervention are either haemodynamically significant shunt fraction (Qp/Qs > 1.5) or echocardiographic signs of right heart dilation or RV volume overload and pulmonary hypertension related symptoms.

Exclusion Criteria:

* Patients with a large stretched Secundum ASD ≥ 36 mm, those with insufficient ASD rims (except the aortic rim), sinus venosus or primum type ASD, irreversible pulmonary hypertension, other associated structural heart diseases, coronary artery disease, LV systolic dysfunction, atrial fibrillation, or hypertension.

Min Age: 11 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study includes two groups: 1. Patients with isolated Secundum ASDs who are referred for possible elective transcatheter closure of the defects. Comparison between the results of the haemodynamic 2D echocardiography derived Strain and Strain Rate imaging procedure will be done as follow:
  a. Echo 1 - performed just before the procedure b. Echo 2 - performed the day after the procedure c. Echo 3 - performed 1-3 months following the procedure
  2. Control group: age and gender-matched healthy subjects are being examined to assess their LV and RV haemodynamic parameters and strain results and compare these data with the study group.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Measuring of the biventricular geometrical changes before and after ASD device closure | 1-3 month
  The LV and RV geometrical changes of the ASD group will be evaluated by using standard 2D Transthoracic Echocardiography before, 24 hours and one month after transcatheter ASD device closure procedure. The geometrical changes include LV and RV dimensions, pressure and wall masses.
Measure change from baseline in the biventricular function of the ASD group | 1-3 month
  Change from baseline in Biventricular systolic function and LV diastolic function of the ASD group will be measured by using 2D Echocardiography (derived Strain, Strain Rate and Tissue Doppler Imaging) at 24 hours and one month after transcatheter ASD device closure procedure.
Measure the biventricular geometry and function of the control group | Baseline
  The control group LV/RV geometry and function values will be evaluated by using 2D Transthoracic Echocardiography.
Measure the relationship between the geometrical and function changes and device size of the ASD group | 1-3 month
  The waist size of the selected device that will be used in transcatheter closure of the ASD will be documented according to the diameter of defect by using Transoesophageal Echocardiography before and during the closure procedure. Then, the relationship between the LV/RV geometrical and function changes after transcatheter closure and the used device size will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Areej AA Tammam Alkhateeb, Msc, Principal Investigator — Assiut University; Alaa M Roushdy, MD,PhD, Principal Investigator — Ain Shams University; Ayman KM Hassan, MD,PhD, Study Chair — Assiut University; Hosam Hasan-Ali, MD, PhD, Study Director — Assiut University; Yehia T Kishk, MD, PhD, Study Director — Assiut University
Locations (2):
- Egypt (2):
  - Assiut University Hospital, Asyut
  - Ain Shams University Hospital, Cairo

REFERENCES:
- [Result] Lange A, Coleman DM, Palka P, Burstow DJ, Wilkinson JL, Godman MJ. Effect of catheter device closure of atrial septal defect on diastolic mitral annular motion. Am J Cardiol. 2003 Jan 1;91(1):104-8. doi: 10.1016/s0002-9149(02)03013-8. No abstract available. PMID 12505587
- [Result] Bussadori C, Oliveira P, Arcidiacono C, Saracino A, Nicolosi E, Negura D, Piazza L, Micheletti A, Chessa M, Butera G, Dua JS, Carminati M. Right and left ventricular strain and strain rate in young adults before and after percutaneous atrial septal defect closure. Echocardiography. 2011 Aug;28(7):730-7. doi: 10.1111/j.1540-8175.2011.01434.x. Epub 2011 May 25. PMID 21615485
- [Result] Balci KG, Balci MM, Aksoy MM, Yilmaz S, Ayturk M, Dogan M, Yeter E, Akdemir R. Remodeling process in right and left ventricle after percutaneous atrial septal defect closure in adult patients. Turk Kardiyol Dern Ars. 2015 Apr;43(3):250-8. doi: 10.5543/tkda.2015.57106. PMID 25905996
- [Result] Wu ET, Akagi T, Taniguchi M, Maruo T, Sakuragi S, Otsuki S, Okamoto Y, Sano S. Differences in right and left ventricular remodeling after transcatheter closure of atrial septal defect among adults. Catheter Cardiovasc Interv. 2007 May 1;69(6):866-71. doi: 10.1002/ccd.21075. PMID 17390329